CLINICAL TRIAL: NCT05816837
Title: Displacement Distance and Stabilization Time for Liver Fiducial Marker
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Peking University Third Hospital (Other)
Responsible Party: Principal Investigator, Qiu Bin, Principal Investigator, Peking University Third Hospital
Other Study IDs: 3D-LVFM-1
Record Dates: First submitted 2023-04-04; First posted 2023-04-18 (Actual); Last update posted 2023-04-18 (Actual); Status verified 2023-04

CONDITIONS: Liver Cancer
Keywords: liver cancer
MeSH Terms: conditions — Liver Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Liver malignant tumor, including liver cancer and liver metastasis, is common in China [1]. Previous studies have shown that cyber-knife stereotactic radiotherapy is effective and safe for locally advanced liver malignancies with improved local tumor control [2]. Real-time tumor tracking in cyber-knife stereotactic radiotherapy is currently used as tumors have respiratory movements [3]. At present, fiducial marker is used to realize the real-time track of tumor [4, 5]. However, the fiducial marker are likely to displacement usually within 7 days after implantation [4, 6, 7]. Therefore, simulated CT are delayed 7 days before the fiducial marker stabilization and significantly extend the radiotherapy planning process, increase the risk of tumor progression. As far as we know, there is no prospective study on the specific displacement distance and duration before the fiducial marker stabilization after implantation. Therefore, the purpose of this study was to study the displacement distance and stabilization time before stereotactic radiotherapy for liver malignant tumors guided by 3D printing template-assisted CT.

1. B.K. Chang, R.D. Timmerman, Stereotactic body radiation therapy: a comprehensive review, Am J Clin Oncol 30 (6) (2007) 637-644.
2. Kato Y, Kamomae T, Kumagai M, Oie Y, Noguchi Y, Okudaira K, et al. Hybrid 3D T1-weighted gradient-echo sequence for fiducial marker detection and tumor delineation via magnetic resonance imaging in liver stereotactic body radiation therapy. 2022;95:9-15.
3. D.K. Bhasin, S.S. Rana, S. Jahagirdar, B. Nagi, Does the pancreas move with respiration? J Gastroenterol Hepatol 21 (9) (2006) 1424-1427.
4. N. Kothary, J.J. Heit, J.D. Louie, W.T. Kuo, B.J. Loo, A. Koong, D.T. Chang, D. Hovsepian, D.Y. Sze, L.V. Hofmann, Safety and efficacy of percutaneous fiducial marker implantation for image-guided radiation therapy, J. Vasc. Interv. Radiol. 20 (2) (2009) 235-239.
5. C.G. Trumm, S.M. Häussler, A. Muacevic, R. Stahl, S. Stintzing, P.M. Paprottka, F. Strobl, T.F. Jakobs, M.F. Reiser, R.T. Hoffmann, CT fluoroscopy-guided percutaneous fiducial marker placement for CyberKnife stereotactic radiosurgery: technical results and complications in 222 consecutive procedures, J. Vasc. Interv. Radiol. 25 (5) (2014) 760-768.
6. Y. Seppenwoolde, W. Wunderink, V.S. Wunderink-van, P. Storchi, R.A. Méndez, B.J. Heijmen, Treatment precision of image-guided liver SBRT using implanted fiducial markers depends on marker-tumour distance, Phys. Med. Biol. 56 (17) (2011) 5445-5468.
7. K. Valentine, T. Cabrera, D. Roberge, Implanting metal fiducials to guide stereotactic liver radiation: McGill experience and review of current devices, techniques and complications, Technol Cancer Res Treat 13 (3) (2014) 253-258.

ELIGIBILITY:
Inclusion Criteria:

1. Ages 18 to 85
2. Single or multiple liver tumors or mass (solid, partially solid)
3. Without taking drugs affecting coagulation and/or platelet aggregation are used; If used, the drug has been discontinued for a sufficient period of time (e.g. 1 week)
4. KPS>60 points, no serious or uncontrolled underlying diseases, clinical evaluation patients can tolerate puncture
5. Planned fiducial marker implantation with applicable puncture path
6. With informed consent.

Exclusion Criteria:

1. Poor organ function
2. The lesion close to blood vessels and intestine, or there is portal vein hypertension and superior vena cava compression, etc., which are expected to have high risks of puncture bleeding and intestinal injury
3. Poor compliance, unable to complete coordination
4. Paticipant who is considered inappropriate or unwilling to participate in this clinical trial for other reasons.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: participant with liver tumors and plan to implant fiducial marker for radiatherapy.
Sampling Method: Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2022-04-20 (Actual); Primary Completion 2024-04-19 (Estimated); Study Completion 2024-04-19 (Estimated)

PRIMARY OUTCOMES:
Displacement distance | Within 1 weeks
  Fiducial marker displacement distance (millimeter) in the liver after implantation

CONTACTS AND LOCATIONS:
Locations (2):
- China (2):
  - Peking University Third Hospital, Beijing, United Kingdom of Great Britain and Northern Ireland
  - Department of Radiation Oncology of Peking university third hospital, Beijing

IPD SHARING:
Plan to Share IPD: Undecided